CLINICAL TRIAL: NCT06153836
Title: Randomized Feasibility Study to Determine the Feasibility of Neurotization of the Nipple Areolar Complex at the Time of Nipple Sparing Mastectomy and Prosthetic Based Reconstruction
Brief Title: Neurotization of the Nipple Areolar Complex to Restore Sensation for Patients With Breast Cancer Undergoing Nipple Sparing Mastectomy and Reconstruction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC230302; NCI-2023-09574 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-004411 (Other: Mayo Clinic Institutional Review Board); MC230302 (Other: Mayo Clinic)
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Carcinoma In Situ | interventions — Mastectomy, Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM I (control) (Active Comparator): Patients undergo standard of care NSM on study.
  Interventions: Other: Questionnaire Administration; Procedure: Subcutaneous Mastectomy
- ARM II (neurotization) (Experimental): Patients undergo neurotization during standard of care NSM on study.
  Interventions: Procedure: Neurotization Procedure; Other: Questionnaire Administration; Procedure: Subcutaneous Mastectomy

INTERVENTIONS:
Procedure: Neurotization Procedure — Undergo placement of nerve graft
  Other Names: Nerve Regeneration Procedure
  Arms: ARM II (neurotization)
Other: Questionnaire Administration — Ancillary studies
Procedure: Subcutaneous Mastectomy — Undergo standard of care NSM
  Other Names: Nipple-Sparing Mastectomy

SUMMARY:
This phase II trial tests the willingness of patients undergoing nipple sparing mastectomy (NSM) to enroll in a randomized study of NSM with or without neurotization of the nipple areolar complex (NAC). This trial also compares patient reported outcomes, including quality of life and breast and NAC sexual functionality, for patients undergoing NSM with or without neurotization of the NAC. NSM is a standard practice option for patients undergoing preventative mastectomy, but many report dissatisfaction with decreased nipple sensation. Neurotization is a surgical technique using a nerve graft in an attempt to restore NAC sensation. Neurotization during NSM and reconstruction may restore NAC sensation and improve quality of life in breast cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine willingness of patients undergoing NSM to enroll in a randomized trial of NSM with or without neurotization.

SECONDARY OBJECTIVES:

I. To compare patient reported outcomes, including quality of life and breast and NAC sexual functionality, for patients undergoing NSM with or without neurotization.

II. To compare NAC sensation at 12 months in patients undergoing NSM with or without neurotization.

III To determine rate of mastectomy skin flap necrosis following NSM via the skin ischemia and necrosis (SKIN) score.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo standard of care NSM on study.

ARM II: Patients undergo neurotization during standard of care NSM on study.

After completion of study intervention, patients are followed at 14 days and at 6, 12 and 24 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Female patients age >= 18
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Planned nipple sparing mastectomy (NSM)
* Ideal NSM candidates would meet the following criteria:

  * Cup size A-C
  * BMI <34
  * Ptosis grade < 2
  * Clinical stage 0 - T2N0
  * Final planned implant volume < 400cc
  * Inframammary or lateral mammary incision
  * Tumor > 0.5cm from the nipple areolar complex (NAC)
  * No prior breast reduction, mastopexy, or periareolar incisions on side of planned NSM
  * No prior breast radiation on side of planned NSM
  * Tumor <0.5cm from NAC (including suspicious calcifications or MRI enhancement)
  * No planned post mastectomy radiation (PMRT)
  * No nicotine use within 4 weeks of surgical date

Exclusion Criteria:

* Planned autologous reconstruction (immediate or delayed)
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2026-11-10 (Estimated); Study Completion 2026-11-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients undergoing nipple sparing mastectomy (NSM) to enroll in a randomized trial of NSM with or without neurotization | Up to 2 years
  Will calculate the proportion of eligible patients who opt to take part in the study. Additionally, will descriptively analyze and report the specific factors that influenced patients' decisions to participate, with the aim of identifying and addressing any obstacles encountered.

SECONDARY OUTCOMES:
Chest physical well-being | At baseline and up to 12 months
  Measured using the BREAST-Q© scored on a 3-point Likert scale where 1=None of the time and 3=All of the time. Higher scores indicate poorer chest physical well-being.
Psychosocial well-being | At baseline and up to 12 months
  Measured using the BREAST-Q© scored on a 5-point Likert scale where 1=None of the time and 5=All of the time. Higher scores indicate poorer psychosocial well-being.
Sexual well-being | At baseline and up to 12 months
  Measured using the BREAST-Q© scored on a 5-point Likert scale where 1=None of the time and 5=All of the time. Higher scores indicate poorer sexual well-being.
Patient reported amount of sensation in nipple areolar complex (NAC) and breast | At baseline and up to 12 months
  Patient reported amount of sensation in nipple areolar complex (NAC) and breast will be will be assessed using a 5-item sensation questionnaire with 5 options to answer each question. Examples of answers include a range from Very unpleasant to Very pleasant or Unimportant to Very Important. Results will be reported descriptively.
Patient reported significance of breast or NAC for sexuality | At baseline and up to 12 months
  Patient reported significance of breast or NAC for sexuality will be assessed using a 5-item Significance of Breast or Nipple Areolar Complex for Sexuality Questionnaire with 5 options to answer each question: Not at all, A little bit, Somewhat, Quite a bit, or Very much. Results will be reported descriptively.
Tactile sensitivity scores | At baseline and up to 12 months
  Measured using Semmes Weinstein monofilament test. Scores will be averaged for each patient across all breast/ NAC measurements and summarized in terms of mean, standard deviation, median, and range. The ordinal score at each of the sites will also be summarized in terms of median and range. Frequency and type of missing data will be summarized.
Incidence of adverse events (AEs) | At 12 months
  AEs will be scored using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) and will be summarized within arms by reporting the number and percentage of patients for each AE. The maximum grade for each type of AEs will be recorded for each patient and frequency tables will be reviewed to determine overall patterns. The frequency and type of solicited AEs experienced in each arm will also be reported.
Mastectomy skin flap necrosis | At 12 months
  Incidence of mastectomy skin flap necrosis will be assessed using the skin ischemia necrosis (SKIN) score, as recorded by clinical staff. Necrosis is defined as any depth SKIN score of C or D and surface area >1.

CONTACTS AND LOCATIONS:
Overall Officials: James W. Jakub, M.D., Principal Investigator — Mayo Clinic; Olivia S. Ho, M.D., M.S., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials